CLINICAL TRIAL: NCT06016751
Title: Relationship Between Intracranial Blood Flow and Peripheral Perfusion in Patients With Craniocerebral Injury Assessed by Doppler Ultrasound and Prognostic Assessment
Brief Title: Relationship Between Intracranial Blood Flow and Peripheral Perfusion in Patients With Craniocerebral Injury
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YLong
Record Dates: First submitted 2023-07-19; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Brain-injury; Intracranial; Blood Vessel, Injury
MeSH Terms: conditions — Brain Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cranial damage: Our study was a prospective observational study which included only a group of patients who were diagnosed with acute craniocerebral injury.

SUMMARY:
Neurocritical care is a major branch in the field of critical care medicine, and more than 50% of the neurocritical care patients in the Tibet Autonomous Region People's Hospital (TARPH) are in neurocritical care, of which cranial damage accounts for about 30%, and paroxysmal sympathetic hyperexcitability syndrome (PSH) after traumatic brain injury（TBI）is a common complication, which affects the cardiorespiratory and cerebral functions to varying degrees, and optimizing the cerebral perfusion and oxygenation supply is the key point in the treatment of TIB, and the maintenance of the cerebral homeostasis and the functional homeostasis is currently an international hotspot for treatment. Maintaining cerebral homeostasis and body function homeostasis is an international hotspot in the treatment of TIB. This study intends to elaborate on the relationship between PSH and Intracranial blood flow in patients with TBI, as well as the effect of anti-stress treatment on Intracranial blood flow. Implementation Patients with brain injury admitted to our department from January 2021 to January 2022 were included. Non-invasive transcranial Doppler ultrasound was applied to measure cerebral blood flow, non-invasive local cerebral oxygen saturation monitor to measure local cerebral oxygen saturation, and an electroencephalography bispectrometer to measure BIS score to quantify the depth of sedation during the experimental process. Bedside ultrasound monitored the right heart function and lung water status, and the data of each monitoring index were monitored and recorded throughout the whole process, and the relationship between concomitant PSH and Intracranial blood flow in TBI patients was found according to the statistical analysis. Ultimately, to achieve the control of TBI complications and improve patient rescue. To expect to achieve the purpose of improving the prognosis of TBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Craniocerebral injury patients;
* The middle cerebral artery blood flow spectrum can be clearly displayed with a bedside TCD;

Exclusion Criteria:

* Age Under 18 years;
* history of cardiovascular disease such as coronary artery disease, heart failure, or atrial fibrillation;
* presence of severe valvular disease or ejection fraction (EF) <30%;
* chronic lung disease;
* chronic liver failure or renal insufficiency;
* persons with co-morbidities of malignant neoplasms;
* persons who had co-morbidities with acute and chronic infectious diseases prior to craniocerebral injuries;
* women who were pregnant and breastfeeding;
* history of psychiatric disorders;
* history of drug abuse or alcohol misuse;
* history of β-blockers;
* co-morbidities with spinal cord injuries; and persons who had died or been discharged from hospital within 1 week of hospitalization or who had not been able to obtain a clear image with ultrasonography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Definite craniocerebral injury, surgically treated and transferred to ICU.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
intracranial blood flow | Day 1,Day 3,Day 5
  Mean intracranial middle cerebral artery blood flow velocity and pulsatility index measured using ultrasound Doppler in enrolled patients.
Paroxysmal sympathetic excitation | Day 1,Day 3,Day 5
  Use of the Paroxysmal Sympathetic Nerve Score to assess paroxysmal sympathoexcitatory performance in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Du, Beijing, Beijing Municipality, China